CLINICAL TRIAL: NCT02681536
Title: Miniflare Versus Long Protocol in Poor Responders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Dina Mohamed Refaat Dakhly, Lecturer of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: FS090216
Record Dates: First submitted 2016-02-09; First posted 2016-02-12 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate; drospirenone and ethinyl estradiol combination; hMG-IBSA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minidose long protocol (Experimental): Down-regulation started on day 20 of the previous cycle by GnRH agonist triptorelin (0.5 µg Decapeptyl; Ferring). On the second day of menstruation, when down regulation was confirmed (as evidenced by endometrial thickness <5 mm and/or E2 levels <50 pg/mL) using transvaginal sonography (TVS) by Voluson 730 Pro (GE, Fairfield, CT) apparatus, gonadotropin (Merional; IBSA) was commenced at an initial dose of 300-450 IU/day for the first 5 days followed by individual adjustment in Gn dose according to ovarian response and the dose of Decapeptyl 50µg/day was continued until day of HCG administration.
  Interventions: Drug: Triptorelin; Drug: HMG
- microdose flare protocol (Experimental): OCPs drospirenone /ethinyl estradiol (Yasmin, BAYER) for not less than 21 days before starting ovarian stimulation, this was followed by 2 days free. Triptorelin (Decapeptyl Ferring Pharmaceuticals, Germany) 0.05 mg/day S.C. was then started daily followed by HMG IM daily (Merional, 75 IU, IBSA) 3 days later. Then the same cycle adjustment was done as the minidose long protocol.
  Interventions: Drug: Triptorelin; Drug: Combined oral contraceptive pills; Drug: HMG

INTERVENTIONS:
Drug: Triptorelin
  Other Names: Decapeptyl
Drug: Combined oral contraceptive pills
  Other Names: Yasmin
  Arms: microdose flare protocol
Drug: HMG
  Other Names: merional

SUMMARY:
The study is performed to compare the outcomes of two stimulation protocols, the minidose long protocol versus the microdose flare protocol in poor responders undergoing IVF/ICSI.

ELIGIBILITY:
Inclusion Criteria:

* poor responder women who fulfilled the criteria defined by the ESHRE consensus in 2011[4]; Poor responder females are those who possess two out of these three criteria: i) Female age ≥40 years; ii) Females who have at least one previous cancelled IVF cycle; iii) POR according to AFC ≤5 or low AMH value.

Exclusion Criteria:

* females with FSH more than 20 IU/L
* females with previous ovarian surgery
* females suffering from causes of infertility other than poor ovarian response, cases with polycystic ovaries syndrome
* females refusing to be enrolled in the study, females with any endocrine disorder such as: diabetes, thyroid
* patients with male factor of infertility.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes retrieved | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dina MR Dakhly, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr el aini hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Siristatidis CS, Yong LN, Maheshwari A, Ray Chaudhuri Bhatta S. Gonadotropin-releasing hormone agonist protocols for pituitary suppression in assisted reproduction. Cochrane Database Syst Rev. 2025 Jan 9;1(1):CD006919. doi: 10.1002/14651858.CD006919.pub5. PMID 39783453